CLINICAL TRIAL: NCT00005657
Title: Immunogenetics of Hepatitis C Virus Infection
Brief Title: Genetics of Hepatitis C Virus Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000125; 00-DK-0125
Record Dates: First submitted 2000-05-06; First posted 2000-05-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-19

CONDITIONS: Hepatitis C; Liver Disease
Keywords: Cytokines; Treatment; Genetic Polymorphism; Chronic Hepatitis C; Mononuclear Cells
MeSH Terms: conditions — Hepatitis C; Liver Diseases; Hepatitis C, Chronic

SUMMARY:
The diverse clinical syndromes associated with hepatitis C underscore the multifactorial and polygenic nature of HCV infection. Both viral and host factors likely contribute to variations in infection outcome, disease susceptibility and progression, and treatment response. This protocol will focus on the immunogenetics of HCV infection. Various candidate genes, most of them related to host immune response in microbial infection, have defined genetic polymorphisms that have been associated with variable manifestations of infections including malaria, tuberculosis, leprosy, AIDS and hepatitis B. In this proposal, we plan to collect peripheral blood mononuclear cells as a source of DNA from approximately 1500 patients with HCV infection, analyze genetic polymorphisms of various candidate genes in association with viral clearance, disease progression or treatment response, and characterize the functional consequences of these polymorphisms in patients with well-defined clinical sequelae of HCV infection. We will also collect blood from patients with other forms of liver diseases (approximately 300) or normal volunteers (approximately 200) as controls. By identifying relevant host factors genetically and investigating their molecular interactions with HCV, we may gain additional insights into HCV pathogenesis and uncover new potential targets for vaccine development and treatment intervention.

DETAILED DESCRIPTION:
The diverse clinical syndromes associated with hepatitis C underscore the multifactorial and polygenic nature of HCV infection. Both viral and host factors likely contribute to variations in infection outcome, disease susceptibility and progression, and treatment response. This protocol will focus on the immunogenetics of HCV infection. Various candidate genes, most of them related to host immune response in microbial infection, have defined genetic polymorphisms that have been associated with variable manifestations of infections including malaria, tuberculosis, leprosy, AIDS and hepatitis B. In this proposal, we plan to collect peripheral blood mononuclear cells as a source of DNA from approximately 1500 patients with HCV infection, analyze genetic polymorphisms of various candidate genes in association with viral clearance, disease progression or treatment response, and characterize the functional consequences of these polymorphisms in patients with well-defined clinical sequelae of HCV infection. We will also collect blood from patients with other forms of liver diseases (approximately 300) or normal volunteers (approximately 200) as controls. By identifying relevant host factors genetically and investigating their molecular interactions with HCV, we may gain additional insights into HCV pathogenesis and uncover new potential targets for vaccine development and treatment intervention.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who have recovered from past HCV exposure (positive anti-HCV but negative HCV viremia and absent liver disease).

Patients with asymptomatic HCV infection (positive anti-HCV and HCV viremia, but persistently normal or minimally elevated ALT and normal or mild disease on liver biopsy).

Patients with active liver disease (positive anti-HCV and HCV viremia, persistently elevated ALT and/or moderate disease on liver biopsy).

Patients with active extrahepatic manifestations of HCV infection (cryoglobulinemia, glomerulonephritis, vasculitis, etc.).

Patients with rapidly progressive, severe liver disease and/or hepatocellular carcinoma.

Patients who have undergone or are undergoing treatment.

Patients from a single-source outbreak of HCV infections (in which the viral factors should be identical and the patients are often from a homogeneous population with less genetic variability).

HCV infected family members and twins.

Patients with other forms of liver disease including HBV infection, primary biliary cirrhosis, autoimmune hepatitis, nonalcoholic steatohepatitis, hemochromatosis, and Wilson's Disease, as well as normal volunteers.

EXCLUSION CRITERIA:

Adult subjects with a Hct of less than 30 or pediatric subjects less than 25 will be excluded.

Children with HCV infection younger than 2 years of age will be excluded.

Unaffected healthy volunteers who are minors are not eligible for this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2000-05-04; Study Completion 2011-04-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Todd JR, West BC, McDonald JC. Human leukocyte antigen and leprosy: study in northern Louisiana and review. Rev Infect Dis. 1990 Jan-Feb;12(1):63-74. doi: 10.1093/clinids/12.1.63. PMID 2300741
- [Background] Hill AV, Allsopp CE, Kwiatkowski D, Anstey NM, Twumasi P, Rowe PA, Bennett S, Brewster D, McMichael AJ, Greenwood BM. Common west African HLA antigens are associated with protection from severe malaria. Nature. 1991 Aug 15;352(6336):595-600. doi: 10.1038/352595a0. PMID 1865923
- [Background] Hill AV. The immunogenetics of human infectious diseases. Annu Rev Immunol. 1998;16:593-617. doi: 10.1146/annurev.immunol.16.1.593. PMID 9597143